CLINICAL TRIAL: NCT04026074
Title: Randomized Controlled Doubleblind Pilot Study Comparing Analgosedation Concepts During Placement of Regional Anaesthesia With Either Fentanyl, Remifentanil, Clonidine, EMLA-Patch or Placebo in Regard of Pain Reduction.
Brief Title: Concepts for Analgosedation During Placement of Regional Anaesthesia Before Operations.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Knee Arthropathy; Hip Arthritis; Fractures, Closed
MeSH Terms: conditions — Fractures, Closed | interventions — Fentanyl; Remifentanil; Clonidine; Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Fentanyl i.v. (intravenously) (Experimental): Patients will be administered the medication and additionally will be treated with placebo salve (skin protection salve)
  Interventions: Drug: Fentanyl; Drug: Placebo salve
- Remifentanil i.v. (Experimental): Patients will be administered the medication and additionally will be treated with placebo salve (skin protection salve)
  Interventions: Drug: Remifentanil; Drug: Placebo salve
- Clonidine i.v. (Experimental): Patients will be administered the medication and additionally will be treated with placebo salve (skin protection salve)
  Interventions: Drug: Clonidine; Drug: Placebo salve
- EMLA salve (Experimental): Patients will be administered the medication (salve) and additionally will be administered i.v. saline as placebo
  Interventions: Drug: EMLA Cream; Drug: Placebo iv
- Placebo (Placebo Comparator): Patients will be administered i.v. placebo (0,9% NaCl) and placebo salve (skin protection salve)
  Interventions: Drug: Placebo iv; Drug: Placebo salve

INTERVENTIONS:
Drug: Fentanyl — Weight adapted drug application
  Arms: Fentanyl i.v. (intravenously)
Drug: Remifentanil — Weight adapted drug application
  Arms: Remifentanil i.v.
Drug: Clonidine — Weight adapted drug application
  Arms: Clonidine i.v.
Drug: EMLA Cream — Salve application on the body part where the regional anaesthesia will be administered
  Arms: EMLA salve
Drug: Placebo iv — i.v. administration of 0,9% NaCl
  Arms: EMLA salve; Placebo
Drug: Placebo salve — Skin protection salve (placebo salve) application on the body part where the regional anaesthesia will be administered
  Arms: Clonidine i.v.; Fentanyl i.v. (intravenously); Placebo; Remifentanil i.v.

SUMMARY:
Aim of the study is to specify the best analgosedation technique during placement of regional anaesthesia from the patients' view.

In this double blind randomized trial the investigators will be testing the application of drugs administered intravenously (fentanyl-bolus, remifentanil-infusion, clonidine-bolus) or transcutaneously (EMLA salve) or placebo (NaCl 0,9% i.v. and skin protection salve).

DETAILED DESCRIPTION:
In this doubleblind randomized pilot trial, patients will receive one of five possible combinations to assess which medication leads to the best medication during placement of regional anaesthesia. This assessement includes NRS, patients' satisfaction and wellbeing. The tested substances will be administered intravenously (fentanyl-bolus, remifentanil-infusion, clonidine-bolus) or transcutaneously (EMLA salve). The fifth combination will be the control group with only placebo medication. We expected to get first information for objectifying analgosedation during placement of regional anaesthesia for the conduction of further studies in this field.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients planed electively for orthopedic surgery

Exclusion Criteria:

* Missing patient's consent
* Intolerance against study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Pain intensity during placement of the regional anaesthesia | 1 day
  Pain assessment during placement of the regional anaesthesia with the Numeric Rating Scale (NRS 1 to 10, with 1=lowest pain score, 10=highest pain score). Lower NRS describes a better outcome.

SECONDARY OUTCOMES:
Patients' wellbeing | 1 day
  Wellbeing assessment during placement of the regional anaesthesia with the anaesthesiological questionnaire (ANP anaesthesiological Questionnaire is a self-rating method for the assessment of postoperative complaints, patient wellbeing and satisfaction. The rating scales from 0 to 3, with 0="none" and 3="strongly"). Higher wellbeing values represent a better outcome.
Complication rate (delirium, allergic reactions, cardiopulmonary decompensation) | Through study completion, an average of 1 day
  Complications on operation day will be recorded and compared between the treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor A Schittek, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Hospital LKH Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
After publication of our results, all data will be made available in respect to the austrian data privacy laws
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of our results, all data will be made available in respect to the austrian data privacy laws. Expected for Summer 2020.
Access Criteria: Research groups interested in the data will be granted access.